CLINICAL TRIAL: NCT06221813
Title: A Phase 1b Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of a Prime-Boost Regimen of Three Dose Levels of PHV02, a Nipah Virus Vaccine Candidate (rVSV-ΔG-EBOV GP-NiVG) in Healthy Adults
Brief Title: Study to Evaluate Safety and Immunogenicity of a Prime-Boost Regimen of rVSV-Nipah Virus Vaccine Candidate PHV02 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Public Health Vaccines LLC (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHV02-C-102
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Nipah Virus Infection
Keywords: live, attenuated vaccine; Nipah virus; PHV02; recombinant vesicular stomatitis virus
MeSH Terms: conditions — Henipavirus Infections | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (first 60 subjects) PHV02 high dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 1 (first 60 subjects) PHV02 medium dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 1 (first 60 subjects) PHV02 low dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 1 (first 60 subjects) Placebo (Placebo Comparator)
  Interventions: Biological: Lactated Ringer's
- Cohort 2 (next 60 subjects) PHV02 high dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 2 (next 60 subjects) PHV02 medium dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 2 (next 60 subjects) PHV02 low dose (Experimental)
  Interventions: Biological: PHV02
- Cohort 2 (next 60 subjects) Placebo (Placebo Comparator)
  Interventions: Biological: Lactated Ringer's

INTERVENTIONS:
Biological: PHV02 — Nipah virus vaccine
  Arms: Cohort 1 (first 60 subjects) PHV02 high dose; Cohort 1 (first 60 subjects) PHV02 low dose; Cohort 1 (first 60 subjects) PHV02 medium dose; Cohort 2 (next 60 subjects) PHV02 high dose; Cohort 2 (next 60 subjects) PHV02 low dose; Cohort 2 (next 60 subjects) PHV02 medium dose
Biological: Lactated Ringer's — Placebo
  Arms: Cohort 1 (first 60 subjects) Placebo; Cohort 2 (next 60 subjects) Placebo

SUMMARY:
The goal of this clinical trial is to test the safety and immunogenicity of PHV02 live, attenuated recombinant vesicular stomatitis virus vaccine expressing the Nipah Virus glycoprotein in healthy adult subjects. The main questions it aims to answer are:

* which doses of PHV02 are safe to administer to and well-tolerated by healthy adult subjects as a 2 dose regimen given 1 month apart?
* what is the immunologic response (Nipah-specific IgG ELISA antibody and neutralizing antibodies) to each dose level after a 2-dose regimen given 1 month apart? Participants will receive 2 intramuscular injections of PHV02 (2x105, 2x106, and 2x107 plaque-forming units [pfu]) or placebo on Day 1 and Day 29 and will be followed for 197 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or non-pregnant, non-lactating females
* Given written informed consent
* No clinically significant health problems
* Negative test for SARS-CoV-2
* Agree to avoid conception through Day 57
* Agree to minimize blood and body fluid exposures to others after vaccination through Day 57
* Agree to avoid exposure to immunocompromised persons after vaccination through Day 57
* Agree to avoid employment in industry involved with livestock after vaccination through Day 57

Exclusion Criteria:

* Prior infection with Nipah virus, related Henipaviruses or Ebola virus
* Prior infection with vesicular stomatitis virus (VSV)
* Received VSV-vectored vaccine or Ebola vaccine
* BMI < 18.5 or ≥ 35
* Healthcare worker with direct physical contact with patients
* Childcare worker in direct contact with children 5 years old or younger
* Household contact who is immunodeficient, or on immunosuppressive medication
* Hands-on food preparation job
* Primary care or treatment of cattle, horses, or swine
* Hepatitis B, hepatitis C, HIV-1, HIV-2, diabetes, atopic dermatitis (eczema), chronic inflammatory disease, autoimmune or autoinflammatory disorder, malignancy, chronic or active neurologic disorder
* History of severe reactions to any vaccine or history of severe allergies
* Receipt of investigational product up to 30 days prior to, or planned receipt within 196 days after randomization, or ongoing participation in another interventional clinical trial.
* Receipt of licensed non-live vaccines within 14 days of planned study immunization (30 days for live vaccines) or planned receipt of non-live or live vaccine within 60 days after first study immunization (30 days after the 2nd vaccination).
* Known allergy to components of PHV02
* Injection sites obscured by tattoos or physical condition
* Significant psychiatric or medical condition or laboratory abnormality on screening
* History of Guillain Barre Syndrome or any chronic or acute neurological disorder
* Alcohol or illicit drug abuse within past 5 years
* Pregnant or lactating female
* Administration of blood or IgG within 120 days preceding study
* History of blood donation within 60 days of study
* Unwilling to undergo diagnostic evaluation of rash (skin biopsy, if indicated) or joint symptoms (arthrocentesis if indicated by joint effusion), in both cases if acceptable to subject
* Elective surgery planned during the study period

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with local injection site and systemic adverse events (AEs) | 14 days after each dose
Percentage of participants with joint related symptoms, rash and unsolicited AEs | 28 days after each dose
Percentage of participants with neurologic AEs | Study Days 1-57
Percentage of participants with medically-attended AEs (MAAEs) and serious AEs (SAEs) | From time of injection through final study visit (Day 197)
Proportion of participants with recombinant vesicular stomatitis virus (rVSV) RNA (Cohort 1 only) in plasma, urine and saliva | From time of injection through Day 43
Proportion of participants who seroconvert compared to Day 1 | Day 29 and Day 57
Geometric mean titers of IgG and ELISA neutralizing antibodies | Day 1, 29, 57

CONTACTS AND LOCATIONS:
Overall Officials: Joan Fusco, PhD, Study Chair — Public Health Vaccines; Thomas P Monath, MD, Study Director — Quigley Biopharma; Gray P Heppner, MD, Study Director — Quigley Biopharma
Locations (3):
- United States (3):
  - Cenexel ACT (Anaheim Clinical Trials), Anaheim, California
  - Cenexel RCA (Research Centers of America), Hollywood, Florida
  - Cenexel JBR (JBR Clinical Research), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monath TP, Nichols R, Feldmann F, Griffin A, Haddock E, Callison J, Meade-White K, Okumura A, Lovaglio J, Hanley PW, Clancy CS, Shaia C, Rida W, Fusco J. Immunological correlates of protection afforded by PHV02 live, attenuated recombinant vesicular stomatitis virus vector vaccine against Nipah virus disease. Front Immunol. 2023 Sep 4;14:1216225. doi: 10.3389/fimmu.2023.1216225. eCollection 2023. PMID 37731485